CLINICAL TRIAL: NCT06681727
Title: Feasibility of Accessible Video Mental Healthcare Triage and Assessment - A Clinical Pilot Study
Brief Title: Feasibility of Accessible Video Mental Healthcare Triage and Assessment
Status: Completed | Type: Observational
Sponsor: Region Stockholm (Other Government)
Collaborators: Karolinska Institutet (Other)
Responsible Party: Sponsor
Other Study IDs: PD pilot
Record Dates: First submitted 2024-11-07; First posted 2024-11-08 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-08

CONDITIONS: Psychiatric Disorders
Keywords: Telepsychiatry; Mental Health Triage; Implementation; Primary care
MeSH Terms: conditions — Mental Disorders | interventions — Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 7 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients belonging to Primary care with help seeking for acute psychiatric symptoms
  Interventions: Other: Accessible Video Mental Healthcare Triage and Assessment (IP)

INTERVENTIONS:
Other: Accessible Video Mental Healthcare Triage and Assessment (IP) — Patients aged 18 years and older who were registered at participating primary care centers were eligible to access the IP through a regional healthcare app. IP comprised a brief digital screening followed by a 45-minute video consultation with a mental health professional. Eligible patients could thereafter schedule appointments at cooperating healthcare centers and clinics through the app used for video consultations.
  Other Names: Immediate psychiatry (IP)

SUMMARY:
This study aims to describe the immediate psychiatry (IP) service, patient population, and patient flow, as well as investigate the experiences, acceptability, and feasibility of the IP triage service implemented in Region Stockholm, Sweden.

Patients aged 18 years and older who were registered at participating primary care centers were eligible to access the IP through a regional healthcare app. IP comprised a brief digital screening followed by a 45-minute video consultation with a mental health professional. The study will employ a mixed methods design with data from medical records, patient surveys, interviews with the IP team, and clinician acceptability questionnaires. The quantitative data will be analyzed via descriptive statistics, and the qualitative data will be analyzed via content analysis.

DETAILED DESCRIPTION:
Study Design, Setting, and Ethical Considerations This pilot study, initiated in May 2022, was conducted at a psychiatric clinic affiliated with Karolinska Huddinge Hospital, in collaboration with eight primary care centers in southern Stockholm, Sweden. Data collection occurred from December 19, 2022, to June 30, 2023. The study was ethically approved by the Swedish Ethical Review Authority (2022-03893-01) and adhered to ethical guidelines. Participants were informed about the study's purpose and procedures, with an option to opt out at any time without affecting their care.

The specific research questions were as follows:

1. How many patients received IP, on the basis of the selected recruitment strategy?
2. What were the subsequent care needs in primary and psychiatric care settings identified for patients after using the service?
3. What were the demographics of participants included in the study, such as age, gender, type of psychiatric problems?
4. How did the participants rate their psychiatric concerns in terms of the type of symptoms, symptom severity, symptom onset, and symptom duration?
5. How did the IP team assess patients' psychiatric symptoms and suicidality?
6. How did the participants rate their satisfaction with the IP?
7. Did patient groups recommended for subsequent care in primary and psychiatric care differ in terms of demographics and clinical aspects explored in C-F?
8. How did the IP team experience their work with the intervention?
9. How did participating primary care centers rate the acceptability of IP?

Recruitment Process Participants were recruited through multiple channels including information on the participating primary healthcare websites, posters, verbal information from healthcare providers, and local advertisements. Recruitment was limited to Swedish speakers due to the app's language and logistical issues with interpreter availability.

Participants Inclusion criteria required participants to be 18 years or older and registered with one of the eight participating primary healthcare centers. No exclusion criteria were applied, enabling the study to include patients with both subclinical and severe psychiatric symptoms.

Intervention and Procedure The Immediate Psychiatry (IP) service was delivered entirely through the "Alltid Öppet" app, which provided patients with a digital pathway to book consultations and complete brief screenings. After consultations, patients were invited to fill out a satisfaction survey. A flowchart of the patient journey was developed to visualize the process. The service was developed through an agile, collaborative approach and monitored weekly by a multidisciplinary team. A detailed service manual was produced, covering protocols for risk assessment, consultation procedures, and patient referrals.

Intake, Screening, and Patient Satisfaction Patients completed a brief psychiatric screening upon registration. After the screening, they could schedule a 45-minute video consultation with a mental health professional, without specific professional matching. Post-consultation, patients were provided with a link to an anonymous satisfaction survey.

Team Organization and Competencies The IP team was multidisciplinary, consisting of psychiatrists, psychologists, psychiatric nurses, a mental health therapist, and administrators. The team had a wide range of experience in general psychiatric care, social psychiatry, and suicide prevention.

Consultation Consultations were guided by a semi-structured interview process adapted for this study. Professionals gathered patient histories, screened for psychiatric symptoms, domestic violence, suicidality, and substance use, and collaboratively developed preliminary care plans with patients.

Clinical Documentation Each consultation was documented in a semi-structured format in the electronic medical record system. Preliminary diagnoses, care plans, suicide risk assessments, and other relevant information, such as experiences of abuse, were recorded following the clinic's standard procedures.

Subsequent Care and Referrals Consultations resulted in referrals to primary or psychiatric care, self-help recommendations, or no further action. Patients were responsible for scheduling follow-up appointments, with support from the healthcare system via the app.

Data Collection and Patient Flow Patient data, including demographic information, preliminary diagnoses, and actions taken, were collected through self-reports and medical records. Patient flow was monitored through the app and medical records.

Screening of Psychiatric Concerns A brief 9-item screening tool was used to assess psychiatric symptoms, history, and current use of medications. This tool was developed to facilitate early information gathering and reduce patient burden during intake.

Medical Records and Data Exports The Operational Support team within Region Stockholm Healthcare provided data exports from medical records, which included patients' demographic information, diagnoses, and suicide risk assessments.

Patient Satisfaction Survey The satisfaction survey utilized a 5-point Likert scale to assess multiple dimensions, including the ease of consultation, staff competence, and likelihood of recommending the service.

IP Team Interviews To capture staff experiences, three semi-structured interviews were conducted with IP team members at the end of the intervention period. These interviews focused on roles, patient interactions, and decision-making processes.

Clinician Acceptability at Primary Care Centers Healthcare professionals who received referred patients were surveyed using the Acceptability of Intervention Measure (AIM) to assess the acceptance and perceived usefulness of the IP service.

Data Analysis Descriptive statistics will be used to summarize patient characteristics. Fisher's Exact Test and the Mann-Whitney U Test will be applied for group comparisons. Missing data will be handled through imputation based on mean values. Qualitative content analysis will be used for interview data, involving systematic coding and theme development.

ELIGIBILITY:
Inclusion criteria:

* Adult patients
* Knowledge of Swedish language
* Access to internet
* Belonging to Primary care in Southwest of Stockholm Region
* Seeking help for acute psychiatric symptoms

Exclusion criteria:

* Younger than 18 years old
* Not meeting inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients belonging to primary care in Southwest of Stockholm who seek help for acute psychiatric symtoms.
Sampling Method: Probability Sample
Enrollment: 172 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Patient characteristics | Study period of 7 months
  Patient characteristics and patient flow Data on patient characteristics were collected through self-reported psychiatric concerns as well as preliminary diagnoses and actions initiated by the IP team, as indicated by information from the medical records. Patient flow was monitored through patient medical records.
Brief screening of psychiatric concerns | Study period of 7 months
  The 9-item brief self-reported screening of psychiatric concerns (Supplement A) was used to gather initial information from patients (patient-rated symptoms and the impact of these symptoms on daily life and relationships via a combination of multiple-choice and open-ended questions.) It assesses a range of psychiatric symptoms, including those related to mood disorders, anxiety disorders, stress-related disorders, obsessive-compulsive disorders, and psychotic disorders. Additionally, it screens for self-harm or suicidal thoughts, psychiatric history, and current use of psychopharmaceuticals. The scale is descriptive without numeric score.

SECONDARY OUTCOMES:
Patients demographics | Pre intervention
  Data exports from medical journals and questionnaires were provided by the operational support team within Region Stockholm Healthcare. The information retrieved from the consultation medical records included patients' legal sex and age
Clinical assessments | Study period of 7 months]
  Data exports from medical journals were provided by the operational support team within Region Stockholm Healthcare. The descriptive information retrieved from the consultation medical records included patients' preliminary diagnoses, suicide risk level, number of historic suicide attempts, and current and planned actions based on the consultation.
Patient satisfaction | Study period of 7 months
  The survey utilized a 5-point Likert scale ranging from 1 ("No, not at all") to 5 ("Yes, completely") to measure various dimensions of patient satisfaction. These dimensions included ease of establishing contact, comfort in sharing health-related experiences, satisfaction with the self-care advice received, perceived effectiveness of the consultation, perceived competence of the staff, respectfulness and considerateness of the treatment, involvement in care or treatment decisions, satisfaction with the choice of receiving clinic for subsequent care, and the likelihood of recommending the service to others. The survey items were based on national and regional Swedish patient surveys used in primary and psychiatric healthcare.
Interviews with the IP Team | Study period of 7 months
  Experiences working with the IP were explored through interviews with the IP team. Three 90-minute semistructured retrospective interviews based on 15 questions were conducted with staff who had provided consultations to patients. The interviews were audio recorded and conducted by a psychologist in training, with experience in interview techniques and who was unaffiliated with the project. These interviews took place during the final month of the intervention period with the three remaining staff members-two mental health nurses and one mental health therapist. The topics covered included healthcare professionals' roles, task management, patient interaction strategies, guiding principles, and decision-making processes.
Clinician acceptability at primary care centers | Study period of 7 months
  The mental and medical healthcare professionals who received referred patients were identified through medical records, contacted by email, and asked to complete the anonymous four-item survey "Acceptability of Intervention Measure" (AIM, Weiner et al., 2017) at the end of the study period. The survey evaluated the receiving clinicians' acceptance of the IP intervention via a five-item Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree), assessing the approval, appeal, personal liking, and general welcoming of the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Lina Martinsson, MD PhD, Principal Investigator — Centre for Psychiatry Research, Dept. Clinical Neuro Science. Karolinska Institute
Locations (2):
- Sweden (2):
  - Psychiatry Southwest, Stockholm
  - Psychiatry Southwest,, Stockholm

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-08-22): https://cdn.clinicaltrials.gov/large-docs/27/NCT06681727/ICF_000.pdf